CLINICAL TRIAL: NCT02583308
Title: Impact of the Subglottic Secretions Drainage on the Tracheal Secretions Colonisation: an Ancillary Study of the DEMETER Trial (NCT02515617)
Brief Title: Impact of the Subglottic Secretions Drainage on the Tracheal Secretions Colonisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Collaborators: Ministry of Health, France (Other Government); University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CHD 053-15
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Ventilator-associated Pneumonia
Keywords: Ventilator-associated pneumonia; Surveillance; Subglottic-secretions; Critically ill patients; Prevention
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Period with endotracheal tubes not allowing SSD (Active Comparator): During this period of the DEMETER study (NCT02515617), patients will be intubated with standard endotracheal tubes not allowing Subglottic Secretions
  Interventions: Device: Endotracheal tubes not allowing SSD
- Period with endotracheal tubes allowing SSD (Experimental): During this period of the DEMETER study (NCT02515617), patients will be intubated with specific endotracheal tubes allowing Subglottic Secretions Drainage
  Interventions: Device: Endotracheal tubes allowing SSD

INTERVENTIONS:
Device: Endotracheal tubes not allowing SSD — In each participating center, a bundle of VAP prevention will be applied: elevate the head of the bed to 30°-45°, regular oral care, manage patients with sedation algorithm, assess readiness to extubate daily, intermittent control of endotracheal tube cuff pressure
  Arms: Period with endotracheal tubes not allowing SSD
Device: Endotracheal tubes allowing SSD — In each participating center, a bundle of VAP prevention will be applied: elevate the head of the bed to 30°-45°, regular oral care, manage patients with sedation algorithm, assess readiness to extubate daily, intermittent control of endotracheal tube cuff pressure.
  In addition, SSD will be realized using a 10 ml syringe at in attending frequency of 2 hours.
  Arms: Period with endotracheal tubes allowing SSD

SUMMARY:
Meta-analysis provide evidence for the benefit of the subglottic secretions drainage (SSD) to reduce the occurrence of Ventilator-Associated Pneumonia (VAP). Nevertheless, the diagnosis of VAP is widely considered as subjective and prone to both false-positive and false negative assignments. In ths way, the impact of SSD remains controversial and its use limited in Intensive Care Units. The DEMETER study assessing the medico-economical impact of the the subglottic secretions drainage (NCT02515617) provides the opportunity to evaluate the dynamics of tracheal colonisation with and without the realisation of SSD. This evaluation would reinforce the results observed during the DEMETER study in considering the adjudicated VAP incidence.

This ancillary study will be performed in 14 centers participating to the DEMETER study

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Invasive mechanical ventilation delivered via an endotracheal tube and expected to be required more than 24 hours
* Intubation performed in units in which the specific endotracheal tube allowing the subglottic secretions drainage (SSD) will be available during the SSD period of the trial
* Information delivered

Exclusion Criteria:

* Previous inclusion in the study
* Patients moribund at the Intensive Care Unit admission
* Pregnant, parturient or breast-feeding woman
* Patient hospitalized without consent and/or deprived of liberty by court's decision
* Patient under guardianship or curators
* Lack of social insurance
* Concomitant inclusion in a trial on VAP prevention
* Patient with no comprehension of the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 896 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of pseudomonas aeruginosa presence in tracheal secretions according to the study group. | Until weaning of mechanical ventilation, an expected average of 10 days

SECONDARY OUTCOMES:
Cumulative incidence of staphylococcus aureus presence in tracheal secretions according to the study group. | Until weaning of mechanical ventilation, an expected average of 10 days
Cumulative incidence of enterobacteria presence in tracheal secretions according to the study group. | Until weaning of mechanical ventilation, an expected average of 10 days
Cumulative incidence of streptococcus pneumoniae presence in tracheal secretions according to the study group. | Until weaning of mechanical ventilation, an expected average of 10 days
Cumulative incidence of haemophilus influenzae presence in tracheal secretions according to the study group. | Until weaning of mechanical ventilation, an expected average of 10 days
Cumulative incidence of stenotrophomonas maltophilia presence in tracheal secretions according to the study group. | Until weaning of mechanical ventilation, an expected average of 10 days
Cumulative incidence of acinetobacter baumannii presence in tracheal secretions according to the study group. | Until weaning of mechanical ventilation, an expected average of 10 days
Cumulative incidence of other non-fermenting gram negative bacilli presence in tracheal secretions according to the study group. | Until weaning of mechanical ventilation, an expected average of 10 days
Cumulative incidence of pseudomonas aeruginosa presence in subglottic secretions during the period with endotracheal tubes allowing SSD. | Until weaning of mechanical ventilation, an expected average of 10 days
Cumulative incidence of staphylococcus aureus presence in subglottic secretions during the period with endotracheal tubes allowing SSD. | Until weaning of mechanical ventilation, an expected average of 10 days
Cumulative incidence of enterobacteria presence in subglottic secretions during the period with endotracheal tubes allowing SSD. | Until weaning of mechanical ventilation, an expected average of 10 days
Cumulative incidence of streptococcus pneumoniae presence in subglottic secretions during the period with endotracheal tubes allowing SSD. | Until weaning of mechanical ventilation, an expected average of 10 days
Cumulative incidence of haemophilus influenzae presence in subglottic secretions during the period with endotracheal tubes allowing SSD. | Until weaning of mechanical ventilation, an expected average of 10 days
Cumulative incidence of stenotrophomonas maltophilia presence in subglottic secretions during the period with endotracheal tubes allowing SSD. | Until weaning of mechanical ventilation, an expected average of 10 days
Cumulative incidence of acinetobacter baumannii presence in subglottic secretions during the period with endotracheal tubes allowing SSD. | Until weaning of mechanical ventilation, an expected average of 10 days
Cumulative incidence of other non-fermenting gram negative bacilli presence in subglottic secretions during the period with endotracheal tubes allowing SSD. | Until weaning of mechanical ventilation, an expected average of 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude LACHERADE, MD, Principal Investigator — CHD VENDEE
Locations (15):
- CHU André Vésale, Montigny-le-Tilleul, Belgium
- France (14):
  - CH Annecy Genevois, Annecy
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre Hospitalier Intercommunal des Portes de l'Oise, Beaumont-sur-Oise
  - Chd Vendee, La Roche-sur-Yon
  - CH Docteur Schaffner, Lens
  - CH de Montauban, Montauban
  - Centre Hospitalier Régional d'Orléans, Orléans
  - CHU Pointe-à-Pitre les Abymes, Pointe à Pitre
  - CHI Poissy Saint Germain, Poissy
  - Centre Hospitalier René Dubos, Pontoise
  - CHU La Réunion, site de Saint Denis de la Réunion, Saint-Denis (Réunion)
  - CH de Saint Nazaire, Saint-Nazaire
  - CHU de Strasbourg Nouvel Hôpital Civil, Strasbourg
  - CHU Tours, site Bretonneau, Tours

REFERENCES:
- [Background] Girou E, Buu-Hoi A, Stephan F, Novara A, Gutmann L, Safar M, Fagon JY. Airway colonisation in long-term mechanically ventilated patients. Effect of semi-recumbent position and continuous subglottic suctioning. Intensive Care Med. 2004 Feb;30(2):225-233. doi: 10.1007/s00134-003-2077-4. Epub 2003 Nov 29. PMID 14647884